CLINICAL TRIAL: NCT01195948
Title: Peptide B27PD (Optiquel®) as Corticosteroid-sparing Therapy for Chronic Non-infectious Uveitis (BOOTS)
Brief Title: Optiquel® as Corticosteroid-sparing Therapy for Chronic Noninfectious Uveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100191; 10-EI-0191 (Other: National Institutes of Health)
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2014-12

CONDITIONS: Uveitis
Keywords: Uveitis; Oral Tolerance
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B27PD 1 mg (Experimental): Participants randomly assigned to the B27PD 1 mg arm were instructed to take the capsule orally three times per week (i.e., Monday, Wednesday and Friday) in the morning, at least four hours after the last meal and at least 30 minutes before the next meal for 24 weeks.
  Interventions: Drug: B27PD
- B27PD 4 mg (Experimental): Participants randomly assigned to the B27PD 4 mg arm were instructed to take the capsule orally three times per week (i.e., Monday, Wednesday and Friday) in the morning, at least four hours after the last meal and at least 30 minutes before the next meal for 24 weeks.
  Interventions: Drug: B27PD
- Placebo (Placebo Comparator): Participants randomly assigned to the placebo arm were instructed to take the capsule orally three times per week (i.e., Monday, Wednesday and Friday) in the morning, at least four hours after the last meal and at least 30 minutes before the next meal for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: B27PD
  Other Names: Optiquel®
  Arms: B27PD 1 mg; B27PD 4 mg
Drug: Placebo — Capsule with no active ingredients to mimic B27PD
  Arms: Placebo

SUMMARY:
Background:

Uveitis is a serious inflammatory condition in which the body's immune system attacks parts of the eye, often causing vision loss. Uveitis treatments involve various drugs that suppress the immune system, but these medicines sometimes do not work or may cause serious side effects. Researchers are interested in developing new treatments for uveitis that are more effective and have fewer side effects.

Optiquel® is an experimental medication being tested for its effectiveness against uveitis. It contains B27PD, a small protein fragment, which is similar to proteins in the parts of the eye being attacked by the immune system. Taking Optiquel® (B27PD) by mouth may induce oral tolerance, in which the immune system is taught to recognize and not attack normal parts of the human body.

Objectives:

To evaluate the safety and effectiveness of B27PD (Optiquel®) as a treatment for uveitis.

Eligibility:

Individuals at least 18 years of age who have had noninfectious uveitis in one or both eyes for at least 3 months, have vision of 20/200 or better in at least one eye, and are taking daily prednisone or an equivalent medication.

Design:

Participants will be screened with a physical examination, medical history, blood and urine tests, and an eye exam.

This study will last a maximum of 52 weeks. During the first 12 weeks of the study, participants will have a study visit every 2 weeks. For the remainder of the study, participants will have a study visit every 4 weeks.

Participants will have frequent blood and urine tests, and will also have eye examinations and special procedures (fluorescein angiography and indocyanine green angiography) to evaluate the effectiveness of the treatment.

Participants will be randomly assigned into one of three groups and will receive either one of two different doses of B27PD or a placebo. During the study, participants will also have their dose of prednisone or other steroid medication reduced.

Participants will take one capsule three times per week on Monday, Wednesday, and Friday, for a total of 24 weeks. Participants may take the capsule with water, but should not consume any other drinks or any kind of food until at least 30 minutes have passed to prevent stomach upset. The capsules should be stored in the refrigerator.

DETAILED DESCRIPTION:
Objective: The objective of this study is to evaluate the safety and efficacy of the peptide B27PD (Optiquel®) as a corticosteroid-sparing agent for chronic non-infectious uveitis in participants receiving oral corticosteroid therapy alone or combined with an immunosuppressive agent in a proof-of-concept clinical trial.

Study Population: Patients with non-infectious uveitis requiring at least 20 mg but no more than 40 mg of oral prednisone, or equipotent dose of alternative corticosteroid medication to maintain a quiescent eye, will be eligible.

Design: In this single center, Phase I/II, double-masked, randomized, placebo-controlled, parallel group treatment study, the safety and efficacy of the peptide B27PD will be investigated in 60 participants with non-infectious uveitis. Initially, 60 participants were to be enrolled; however, due to lack of efficacy, only 31 participants were enrolled. Eligible participants will be randomized to one of three treatment groups: 1 mg B27PD, 4 mg B27PD or placebo, to be taken three times per week for 24 weeks. All remaining participants will be followed through a common termination date. The common termination date will be established once the last enrolled participant reaches his/her Week 28 visit (four weeks following his/her last investigational treatment).The time to recurrence of uveitis in either eye occurring in the 52 weeks following the initial dosing will be evaluated in each treatment group. Recurrence will be defined as an increase in anterior chamber cells and/or vitreous haze of at least 2 steps [using the Standardization of Uveitis Nomenclature (SUN) grading system]. Ophthalmic examinations to assess uveitis will include visual acuity, intraocular pressure (IOP), slit lamp biomicroscopy, ophthalmoscopy, optical coherence tomography (OCT) and fluorescein angiography.

Outcome Measures: The primary outcome variable is the time to recurrence of uveitis activity in participants of each treatment group, during or after tapering of oral prednisone to a dose of 7.5 mg/day, or equipotent dose of alternative corticosteroid medication. Secondary efficacy outcome variables include the proportion of participants determined to be a Treatment Failure, defined as recurrence (or flare) of uveitis (at least a 2-step increase using the SUN grading system) or a drop in visual acuity of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters at 24 and 52 weeks. Other secondary efficacy outcomes include the reduction in exposure to corticosteroid as measured by the area under the dose-time curve, and changes in best-corrected visual acuity (BCVA), fluorescein angiography, fundus autofluorescence and high-speed indocyanine green angiography (HS-ICG). Ocular safety measurements include intraocular pressure (IOP) and optical coherence tomography (OCT) for confirmation of suspected macular edema. Systemic safety variables include adverse events, clinical blood chemistry and hematology, urinalysis, vital signs, weight and medical evaluation at baseline and at the end of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant must be 18 years of age or older.
* Participant must be able to understand the informed consent process and sign the informed consent form.
* Participant has been diagnosed with non-infectious unilateral or bilateral uveitis for at least three months. Participants who were diagnosed more than a year prior to enrollment must have had a recurrence in ocular inflammation within the past year.
* Participant must be receiving a current treatment with prednisone between 20 to 40 mg/day (or an equipotent dose of an alternative corticosteroid). Participants who are on a regimen of no more than one anti-metabolite inhibitor at the time of randomization (e.g., azathioprine, methotrexate, mycophenolate) in addition to the prednisone may be enrolled and are allowed to continue the anti-metabolite.
* The participant's uveitis must be controlled in eligible eyes, quiescent eyes [anterior chamber cells and vitreous haze Standardization of Uveitis Nomenclature (SUN) grade of 0].
* The participant's eligible eye(s) is able to be evaluated for activity of disease both biomicroscopically and ophthalmoscopically.
* The participant's baseline intraocular pressure must be > 5 mmHg and ≤ to 30 mmHg in both eyes. Concurrent use of intraocular pressure-lowering medication and/or prior glaucoma surgery is acceptable.
* Participant has best-corrected distance visual acuity in the better seeing eye of 20/200 or better [≥ 34 Early Treatment Diabetic Retinopathy Study (ETDRS) letters].
* Female participants of childbearing potential must not be pregnant or lactating and must be willing to undergo serum pregnancy tests throughout the study.
* Women of childbearing potential must agree to use reliable methods of contraception while receiving the study medication and for 6 weeks following the last administration. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods with spermicide (diaphragm with spermicide, condom with spermicide) or surgical sterilization (hysterectomy, tubal ligation or partner with vasectomy).

EXCLUSION CRITERIA:

* Participant has a non-iatrogenic immunodeficiency state [e.g., Human Immunodeficiency Virus (HIV) infection or congenital immunodeficiency].
* Participant had intraocular surgery or intraocular injection within three months prior to randomization.
* Participant is expected to have an elective ocular surgery or intraocular injection during the study period.
* Participant is using systemic corticosteroid therapy for a non-ocular disease or non-ocular organ involvement.
* Participant has a history or diagnosis of Behcet's disease.
* Participant has a clinically suspected and/or confirmed central nervous system or ocular lymphoma.
* Participant has an active systemic infectious disease or malignancy that requires treatment.
* Participant has a known chronic disease or condition of the gastrointestinal system that may interfere wih the absorption of the investigational product as determined by the investigator (e.g., active hepatitis, chronic diarrhea, inflammatory bowel disease, Crohn's disease, ulcerative colitis, celiac disease, diverticulosis or diverticulitis).
* Participant has two or more food allergies.
* Participant has an implant containing anti-inflammatory, immunosuppressive or antiviral drugs, unless a period 50% longer than the anticipated duration of effect of the implant has elapsed.
* Participant received periocular corticosteroid injections within 4 months prior to randomization or is expected to need periocular corticosteroid injections during the study duration.
* Participant received treatment with infliximab, etanercept, adalimumab, interferon, cyclosporine, tacrolimus, sirolimus, within two weeks prior to randomization.
* Participant received cytotoxic therapy (e.g., cyclophosphamide) within six months prior to randomization.
* Participants for whom, in the physician's opinion, any of the protocol procedures may pose a special risk not outweighed by the potential benefits of participating in the study.
* Participant who is unlikely to comply with the study protocol or who is likely to be moving or lost to follow-up.
* Participant who is currently enrolled or has been participating in any other investigative therapeutic clinical trial during the three months prior to randomization.
* Participant has a known need for a colonoscopy or surgery of the gastrointestinal tract during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Nussenblatt, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barnett ML, Kremer JM, St Clair EW, Clegg DO, Furst D, Weisman M, Fletcher MJ, Chasan-Taber S, Finger E, Morales A, Le CH, Trentham DE. Treatment of rheumatoid arthritis with oral type II collagen. Results of a multicenter, double-blind, placebo-controlled trial. Arthritis Rheum. 1998 Feb;41(2):290-7. doi: 10.1002/1529-0131(199802)41:23.0.CO;2-R. PMID 9485087
- [Background] Dandona L, Dandona R, John RK, McCarty CA, Rao GN. Population based assessment of uveitis in an urban population in southern India. Br J Ophthalmol. 2000 Jul;84(7):706-9. doi: 10.1136/bjo.84.7.706. PMID 10873978
- [Derived] Levy RA, de Andrade FA, Foeldvari I. Cutting-edge issues in autoimmune uveitis. Clin Rev Allergy Immunol. 2011 Oct;41(2):214-23. doi: 10.1007/s12016-011-8267-x. PMID 21913066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Started | 10 | 10 | 11
Week 24 | 10 | 10 | 10
Completed | 10 | 9 | 9
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11.8) | 43 (14.7) | 43 (15.6) | 45 (14.0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 11 | 31
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 8 | 20
  Male | 3 | 5 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome is the Time to Recurrence of Uveitis in Participants of Each Treatment Group, During or After Tapering of Oral Prednisone to a Dose of 7.5 mg/Day, or Equipotent Dose of Alternative Corticosteroid Medication.
Description: Recurrence (or flare) is defined as an anterior chamber cells and/or vitreous haze grading of ≥ 2+ using the Standardization of Uveitis Nomenclature (SUN) grading system.
  The time to this event is defined as the time from randomization to recurrence, loss to follow-up or end of study, whichever comes first. Participants that do not present with disease recurrence will be censored at the time of the last disease evaluation.
Time Frame: Time from randomization to recurrence, loss to follow-up, or end of study, up to 52 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- B27PD 1 mg: Participants randomly assigned to the B27PD 1 mg arm were instructed to take the capsule orally three times per week (i.e., Monday, Wednesday and Friday) in the morning, at least four hours after the last meal and at least 30 minutes before the next meal for 24 weeks.
  B27PD
- B27PD 4 mg: Participants randomly assigned to the B27PD 4 mg arm were instructed to take the capsule orally three times per week (i.e., Monday, Wednesday and Friday) in the morning, at least four hours after the last meal and at least 30 minutes before the next meal for 24 weeks.
  B27PD
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 11
weeks | 52 [52.00 to 52.00] | 52 [28.29 to 52.00] | 45 [10.00 to 52.00]

2. Secondary Outcome: Proportion of Participants Determined to be a Treatment Failure, Defined as Recurrent (or Flare) of Uveitis or a Drop in Visual Acuity of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) Letters
Description: Recurrent (or flare) of uveitis is defined as at least a 2-step increase in anterior chamber cells and/or vitreous haze using the Standardization of Uveitis Nomenclature (SUN) grading system
Time Frame: Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Number; unit: participants
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 1 | 2 | 2

3. Secondary Outcome: Proportion of Participants Determined to be a Treatment Failure, Defined as Recurrent (or Flare) of Uveitis or a Drop in Visual Acuity of ≥ 15 Early Treatment Diabetic Retinopathy Study (ETDRS) Letters
Description: as for outcome 2
Time Frame: Week 52
Population: Twenty-five (25) participants completed Week 52. Three completed prior to Week 52 as a result of early study closure (1/group), two placebo participants and one 4 mg participant were lost to follow-up at Weeks 10, 44 and 28, respectively.
Measure: Number; unit: participants
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 9 | 8 | 8
participants | 1 | 3 | 3

4. Secondary Outcome: Mean Change in Best-Corrected Visual Acuity (BCVA) in Right Eye (OD) at Week 24 Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Mean (Full Range); unit: ETDRS letters
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ETDRS letters | 1.50 [-2.00 to 7.00] | 2.10 [-3.00 to 6.00] | 2.80 [-3.00 to 12.00]

5. Secondary Outcome: Mean Change in Best-Corrected Visual Acuity (BCVA) in Left Eye (OS) at Week 24 Compared to Baseline
Description: as for outcome 4
Time Frame: Baseline and Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Mean (Full Range); unit: ETDRS letters
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
ETDRS letters | 2.80 [-5.00 to 8.00] | 2.00 [-5.00 to 5.00] | 0.50 [-4.00 to 5.00]

6. Secondary Outcome: Number of Participants Presenting No Change in Retinal Vessel Leakage Observed by Fluorescein Angiography (FA) at Week 24 Compared to Baseline
Time Frame: Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Number; unit: participants
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 9 | 9 | 7

7. Secondary Outcome: Number of Participants Presenting No Change in Autofluorescence Patterns as Observed on Fundus Autofluorescence (FAF) at Week 24 Compared to Baseline
Time Frame: Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Number; unit: participants
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 10 | 10 | 9

8. Secondary Outcome: Reduction in Exposure to Corticosteroid as Measured by the Area Under the Dose-time Curve.
Description: This outcome was not analyzed as no data was collected at Week 24.
Time Frame: Week 24
Population: This outcome was not analyzed as no data was collected at Week 24.
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Changes in High-speed Indocyanine Green Angiography (HS-ICG)
Time Frame: Week 24
Population: Thirty (30) participants completed Week 24. One placebo participant was lost to follow-up at Week 10.
Measure: Number; unit: participants
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants
  Increase | 0 | 1 | 0
  Decrease | 0 | 2 | 0
  No change | 10 | 7 | 10

ADVERSE EVENTS:
Time Frame: Maximum of 52 weeks
Arm/Group | B27PD 1 mg | B27PD 4 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B27PD 1 mg (N=10) | B27PD 4 mg (N=10) | Placebo (N=11)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (3) | 2 (2)
Blood urine (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 2 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Creatine urine increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Dental operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Diastolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 2 (4)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eye pruritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin urine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 2 (3)
Heart rate increased (Investigations) | 1 (2) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 4 (4) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (6) | 2 (3) | 4 (5)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscoloskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 1 (1)
Red blood cells urine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 1 (1) | 1 (1)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vulvovaginal pruritis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
White blood cells urine (Investigations) | 0 (0) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pupils unequal (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The protocol was completed early due to lack of efficacy. The Data Safety Monitoring Committee (DSMC), along with the PI, reviewed an interim data report and agreed that Optiquel® was not efficacious and did not cause a proliferative response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes